CLINICAL TRIAL: NCT00620386
Title: Comparing Intubating Conditions and Hemodynamic Changes Between Macintosh Laryngoscopy and Bonfils Fibrescope During Endotracheal Intubation Without Neuromuscular Blockade
Brief Title: Endotracheal Intubation Using Bonfils Fibrescope Without Neuromuscular Blockade
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Endotracheal Intubation; Hemodynamics; Neuromuscular Blockade
Keywords: Intubating conditions; Bonfils intubation fiberscope; Macintosh laryngoscope; neuromuscular blockade

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intubation with Bonfils intubating fiberscope
  Interventions: Device: Bonfils
- 2 (Active Comparator): Intubation with Macintosh laryngoscopy
  Interventions: Device: Macintosh

INTERVENTIONS:
Device: Bonfils — Endotracheal intubation using Bonfils Intubating Fiberscope
  Arms: 1
Device: Macintosh — Endotracheal intubation using Macintosh laryngoscopy
  Arms: 2

SUMMARY:
We studied intubating conditions and hemodynamic changes during endotracheal intubation employing either Bonfils intubating fiberscope or the conventional Macintosh laryngoscopy in 80 healthy patients candidates for elective surgery requiring endotracheal intubation. We omitted neuromuscular blocking drugs from the induction regimen.

DETAILED DESCRIPTION:
BACKGROUND:

Neuromuscular blocking drugs (NMBDs) are believed to be the dominating antigens causing bronchospasm and anaphylaxis during anaesthesia. Avoidance of these drugs, however, renders compromised intubating conditions and higher morbidity with conventional Macintosh laryngoscopy. Thus, we compared Macintosh laryngoscopy with Bonfils intubation fibrescope without administering NMBDs.

METHODS:

Eighty male and female patients scheduled for elective surgery, aged 15 to 60 years, ASA class II or I, non-obese, with lower risk for difficult intubation were enrolled in this study. They were randomly allocated into the Bonfils group or the Macintosh group (40 each). Following adequate hydration and preoxygenation, midazolam 0.05 mg kg-1 was administered, followed by alfentanil 20 µg kg-1, lidocaine 1.5 mg kg-1, and propofol 2 mg kg-1 intravenously. Tracheal intubation was then carried out using Bonfils intubation fibrescope (Bonfils group) or employing conventional Macintosh laryngoscopy (Macintosh group). The primary outcome measure was the intubating condition, with mean arterial blood pressure and heart rate as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status was class I or II
* body mass index (BMI) < 30
* ability to assume the 'sniffing' position

Exclusion Criteria:

* smokers
* drug users
* pregnant
* expected to present difficult intubation
* history of oesophageal reflux
* any systemic or airway disease
* known allergy to the protocol medications

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
intubating conditions | 7 months

SECONDARY OUTCOMES:
mean arterial pressure (MAP) | 7 months
heart rate (HR) | 7 months
Pulse Oxygen Saturation (SpO2) | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Reza Shariat Moharari, MD, Study Director — Tehran University of Medical Sciences; Eiman Rahimi, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Sina Hospital, Tehran, Tehran Province, Iran